CLINICAL TRIAL: NCT07403136
Title: An Open-Label, Two-Cohort Exploratory Phase II Study of Vebrekotuzumab With or Without PD-1 Inhibitor Immunotherapy in Patients With Advanced Esophageal Squamous Cell Carcinoma Refractory to First-Line Therapy
Brief Title: Vebrekotuzumab ± Anti-PD-1 in Pretreated Advanced ESCC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Kuai Le Zhao, MD, Chief physician, Fudan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESO-Shanghai29
Record Dates: First submitted 2026-01-05; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: Esophageal Squamous Cell Carcinoma; Antibody-drug conjugate; Second-line
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vebrekotuzumab+PD-1 (Experimental): Vebrekotuzumab in combination with an immune checkpoint inhibitor.
  Interventions: Drug: Vebrekotuzumab; Drug: PD-1 antibody
- Vebrekotuzumab (Experimental): Vebrekotuzumab monotherapy.
  Interventions: Drug: Vebrekotuzumab

INTERVENTIONS:
Drug: Vebrekotuzumab — This two-cohort study investigates the novel combination of vebrekotuzumab (an EGFR-targeting ADC) with a PD-1 inhibitor versus vebrekotuzumab monotherapy in patients with advanced ESCC refractory to first-line therapy. It uniquely provides a head-to-head comparison to evaluate the synergistic potential of combining targeted cytotoxicity with immune checkpoint blockade in this specific, treatment-resistant population.
Drug: PD-1 antibody — The PD-1 inhibitor (e.g., pembrolizumab) will be used exclusively in Cohort 1 in combination with vebrekotuzumab. This combination is designed to simultaneously deliver targeted cytotoxicity and immune checkpoint blockade, exploring their potential synergy in patients with advanced ESCC who have progressed after first-line therapy.
  Arms: Vebrekotuzumab+PD-1

SUMMARY:
This study will test a new potential treatment for advanced esophageal squamous cell cancer (ESCC) for patients whose initial treatment has stopped working. Currently, the standard second-line treatment for this cancer is PD-1 inhibitors or chemotherapy alone, which is not very effective, allowing the cancer to grow again after just 1.6 to 3.4 months on average. Therefore, there is a strong need for more effective therapies.

The new treatment is a type of drug called an antibody-drug conjugate (ADC). It is designed to target a specific protein called EGFR, which is found in high amounts on the surface of 50-70% of ESCC cancer cells and is linked to a poorer outlook for patients. This ADC works like a targeted delivery system: an antibody guides a powerful cell-killing drug directly to the cancer cells, aiming to destroy them while reducing harm to healthy cells. Although other drugs targeting EGFR have not successfully improved survival for ESCC patients, this new ADC offers a different and promising approach.

The main goal of this study is to find out if this new EGFR-targeting ADC is effective in helping patients with advanced ESCC live longer without their cancer getting worse.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to voluntarily sign the informed consent form and comply with the protocol requirements.
2. Age ≥18 years on the day of signing the informed consent form, regardless of gender.
3. Life expectancy ≥12 weeks.
4. Patients with histologically confirmed advanced recurrent or metastatic esophageal squamous cell carcinoma (ESCC) and immunohistochemistry (IHC) confirmed positive epidermal growth factor receptor (EGFR) expression (IHC 1+, 2+, or 3+).
5. Have experienced disease progression or intolerability after receiving at least one prior line of systemic therapy, which must have included an immune checkpoint inhibitor (e.g., anti-PD-1/PD-L1 antibody).
6. The patient must be able to provide a tumor tissue sample (paraffin block, paraffin-embedded sections, or fresh tissue sections) from the primary or metastatic site for pathological testing. Archived tumor tissue from the most recent treatment should be used. If archived tissue is unavailable, a new biopsy must be performed.
7. Must have radiographic evidence of disease progression confirmed by the investigator during or after the last treatment regimen. At baseline, there must be at least one measurable extracranial lesion per RECIST 1.1 criteria (longest diameter ≥10 mm on CT scan, or for lymph nodes, short axis ≥15 mm). The measurable lesion should not have been previously irradiated, unless it is within a prior radiation field or was previously treated locally and has documented progression.
8. All adverse events (AEs) from prior anti-tumor therapy have resolved to ≤ Grade 1 per the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 5.0 (except for alopecia, non-clinically significant or asymptomatic laboratory abnormalities).
9. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1 within 7 days prior to the first dose.
10. No serious cardiac dysfunction, with left ventricular ejection fraction (LVEF) ≥50% confirmed by echocardiography or MUGA scan within 28 days prior to the first dose.
11. Adequate organ function within 7 days prior to the first dose, as defined by:

    * Bone marrow: Absolute neutrophil count (ANC) ≥1.5 × 10⁹/L; platelet count ≥100 × 10⁹/L; hemoglobin ≥90 g/L. Patient must not have received any blood transfusion or blood component therapy within 14 days prior to the first dose, nor any biologic response modifiers (e.g., G-CSF, erythropoietin) within 7 days prior to the first dose.
    * Liver: For patients without liver metastases: total bilirubin (TBIL) ≤1.5 × upper limit of normal (ULN); alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 × ULN. For patients with liver metastases: TBIL ≤1.5 × ULN; ALT and AST ≤5 × ULN.
    * Kidney: Serum creatinine (Cr) ≤1.5 × ULN, or calculated creatinine clearance (Cockcroft-Gault formula) ≥50 mL/min.
    * Coagulation: International normalized ratio (INR) ≤1.5 × ULN and activated partial thromboplastin time (aPTT) ≤1.5 × ULN (unless the patient is receiving therapeutic anticoagulation).
12. Male patients with reproductive potential and female patients of childbearing potential must be willing to use effective contraception from signing the ICF until 6 months after the last dose of the study drug. Women of childbearing potential include premenopausal women and women within 2 years of menopause onset. A negative serum pregnancy test result must be confirmed for women of childbearing potential within ≤7 days prior to the first study drug dose.

Exclusion Criteria:

1. History of other primary malignancies. Note: Except for adequately treated basal cell carcinoma of the skin, superficial bladder cancer, squamous cell carcinoma of the skin, or carcinoma in situ of the cervix; or patients with other malignancies who have undergone curative treatment and have been disease-free for ≥5 years may be enrolled.
2. Untreated or unstable parenchymal brain metastases, spinal cord compression, carcinomatous meningitis, or leptomeningeal disease.

   Note: Patients who have received local therapy for brain metastases may be enrolled if brain imaging shows stability for at least 28 days prior to the first dose, with no evidence of cerebral edema, and no requirement for corticosteroid therapy.
3. Presence of uncontrolled third-space fluid (e.g., significant ascites, pleural effusion, or pericardial effusion) that cannot be managed by drainage or other methods. Patients who required drainage to control third-space fluid within 14 days prior to the first dose are excluded.
4. Any severe or uncontrolled systemic disease, in the investigator's judgment, including poorly controlled hypertension (systolic blood pressure >160 mmHg or diastolic blood pressure >100 mmHg), poorly controlled diabetes mellitus, or active bleeding signs, etc.
5. Poorly controlled cardiac disease, including heart failure of New York Heart Association (NYHA) class ≥II, unstable angina, myocardial infarction within the past year, clinically significant supraventricular or ventricular arrhythmia requiring treatment, or long QT syndrome, e.g., QTcF >450 ms (male) or QTcF >470 ms (female).
6. Evidence of active infection, including Hepatitis B (HBsAg positive AND HBV DNA ≥2000 IU/mL, excluding drug-induced or other causes of hepatitis), Hepatitis C (anti-HCV antibody positive AND HCV RNA above the lower limit of detection), or human immunodeficiency virus (HIV) infection; or uncontrolled active bacterial, viral, fungal, rickettsial, or parasitic infections, unless treated and resolved prior to study drug administration.
7. History of hypersensitivity to any component of vebrekotuzumab (histidine, histidine hydrochloride, sucrose, mannitol, polysorbate 80) OR history of ≥Grade 3 hypersensitivity reactions to macromolecular protein agents/monoclonal antibodies.
8. History of primary immunodeficiency or active autoimmune disease requiring systemic immunosuppressive therapy or systemic corticosteroid therapy (at doses ≥10 mg/day prednisone or equivalent) within 2 weeks prior to enrollment.

   Note: Patients with type I diabetes mellitus, hypothyroidism managed with stable hormone replacement therapy (including that caused by autoimmune thyroid disease), psoriasis not requiring systemic therapy, or vitiligo may be enrolled.
9. History of or concurrent interstitial lung disease, radiation pneumonitis, severe chronic obstructive pulmonary disease, severe pulmonary insufficiency, symptomatic bronchospasm, etc.
10. Female patients who are pregnant (positive serum pregnancy test), breastfeeding, or unwilling to use adequate contraception during the study period and for 6 months after the last dose of study drug.
11. Any other condition that, in the investigator's opinion, would make the patient unsuitable for participation in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | At the end of every 2 cycles (each cycle is 21 days)
  ORR is defined as the proportion of subjects in the trial who achieved a confirmed complete response (CR) or partial response (PR) as assessed by the investigator according to RECIST v1.1 and iRECIST criteria.

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | At the end of every 2 cycles (each cycle is 21 days)
  DCR is defined as the proportion of subjects achieving complete response (CR), partial response (PR), or stable disease (SD) sustained for at least 5 weeks from the first dose, as assessed by the Independent Review Committee (IRC) per RECIST v1.1 and iRECIST criteria.
Progression-Free Survival (PFS) | The time from the first dose of study treatment until disease progression or death from any cause, whichever occurs first, assessed up to 24 months
  PFS is defined as the time from the first dose of study treatment until disease progression or death from any cause, whichever occurs first.
Overall survival (OS) | The time from the first dose of study treatment until death from any cause, assessed up to 24 months.
  OS is defined as the time from the first dose of study treatment until death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No